CLINICAL TRIAL: NCT04648202
Title: A Phase 1/1b Open-Label Study to Evaluate the Safety and Antitumor Activity of FS120, an OX40/CD137 Bispecific Antibody, Alone and in Combination With Pembrolizumab, in Subjects With Advanced Malignancies
Brief Title: FS120 Phase 1/1b Study in Patients With Advanced Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: invoX Pharma Limited (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FS120-19101; 2021-002820-19 (EudraCT Number); MK-3475-C82 (Other: Merck Sharp & Dohme LLC); KEYNOTE-C82 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2024-10

CONDITIONS: Advanced Cancer; Metastatic Cancer
Keywords: Immuno-oncology; Bispecific antibody; Dose escalation; Cohort expansion; OX40; CD137 (4-1BB); invoX; Pembrolizumab; PD-1
MeSH Terms: conditions — Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FS120 (Experimental): Open-label study where FS120 will be administered as monotherapy or in combination with pembrolizumab in dose escalation and expansion cohorts
  Interventions: Drug: FS120

INTERVENTIONS:
Drug: FS120 — Dosing of participants with FS120 or the combination pembrolizumab will occur intravenously (IV), at a fixed dose in treatment cycles once every 4 weeks (Q4W) or once every 3 weeks (Q3W) until confirmed progressive disease (CPD)/immune-confirmed progressive disease (iCPD) or unacceptable toxicity.
  Other Names: Pembrolizumab (KEYTRUDA®)

SUMMARY:
This is a Phase 1/1b, multicenter, open label study to evaluate the Safety and Antitumor Activity of FS120, an OX40/CD137 Bispecific Antibody, Alone and in Combination with Pembrolizumab, in Subjects with Advanced Malignancies

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease
* Eastern Cooperative Oncology Group Performance Status 0-1.
* Highly effective contraception if risk of conception exists
* A female subject is eligible if not pregnant, not breastfeeding, not a woman of childbearing potential (WOCBP) or is a WOCBP that uses highly effective contraception
* Subjects with HIV who are healthy and how a low risk of acquired immunodeficiency syndrome related outcomes
* For combination part: Subjects must have histologically confirmed locally advanced, unresectable or metastatic solid tumours where there is regulatory approval for use of pembrolizumab as a monotherapy agent

Exclusion Criteria:

* Prior systemic anticancer therapy within 28 days or 5- half-lives, whichever is shorter, before the first dose of study drug.
* Prior therapy with any OX40 agonist, CD137 (4-1BB) agonist, CD40 agonist, GITR, or CD27 targeting therapy (single agent or combination).
* Prior radiotherapy within 2 weeks of start of study treatment.
* HIV infected participants with a history of Kaposi sarcoma and/or Multicentric Castleman Disease.
* Uncontrolled central nervous system (CNS) metastases and/or carcinomatous meningitis, primary CNS tumours, or solid tumours with CNS metastases as the only measurable disease.
* Prior history of any grade ≥3 immune-related AE (irAE) that has not improved to grade ≤1; any grade ≥3 irAE that resulted in discontinuation of treatment, significant (grade ≥3 NCI CTCAE Version 5.0) treatment-related cytokine release syndrome.
* Use of immunosuppressive agents, hypersensitivity or intolerance to monoclonal antibodies or their excipients, persistent grade ≥1 NCI CTCAE Version 5 toxicity related to prior therapy or any condition that would significantly impair and/or prohibit the participant's participation in the study, as per the investigator's judgement.
* Vaccination with a live vaccine within 30 days before first dose of study drug.
* Participants with a known additional malignancy that is progressing or has required active treatment in the past 3 years.
* Participants with severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity, and duration of adverse events (AEs), serious adverse events (SAEs) and dose limiting toxicities (DLTs) | 24 months
  Safety and tolerability will be evaluated by collection of AEs, SAEs and DLTs according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0.
Determination of a maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) | 24 months
  Toxicity will be evaluated according to the NCI CTCAE Version 5.0.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (4):
  - Yale University, New Haven, Connecticut
  - MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
- Spain (5):
  - NEXT Oncology, Hospital Quironsalud Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia